CLINICAL TRIAL: NCT03681639
Title: A Multi-Centre, Prospective Study to Obtain Survival and Clinical Outcome Data on the Zimmer Hip Resurfacing System Utilising the Metasul Monoblock Component™ Cup in a Hip Resurfacing Application With the Durom® Hip Resurfacing Femoral Component.
Brief Title: Metasul Monoblock Component™ Cup in a Hip Resurfacing Application With the Durom® Hip Resurfacing Femoral Component
Acronym: MMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-H00
Record Dates: First submitted 2018-09-13; First posted 2018-09-24 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-10

CONDITIONS: Avascular Necrosis of Hip; Osteoarthritis, Hip; Rheumatoid Arthritis; Inflammatory Arthritis; Post-traumatic; Arthrosis
Keywords: Hip resurfacing; Medical Device; Safety; Hip prosthesis
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis, Rheumatoid; Arthritis; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients who received Metasul Monoblock in hip resurfacing (Experimental): Patients who received the Zimmer Hip Resurfacing System utilising the Metasul Monoblock Component Cup in a Hip Resurfacing Application with the Durom Hip Resurfacing Femoral Component and whose Serum metal ion levels is being measured.
  Interventions: Diagnostic Test: Serum Metal ion levels determined to monitor changes in chromium and cobalt levels

INTERVENTIONS:
Diagnostic Test: Serum Metal ion levels determined to monitor changes in chromium and cobalt levels — Analyses was performed pre-operatively, 6 months, 1 year, 2 years and 5 years post-operatively for all study subjects enrolled in this study, as well as, all revision study subjects receiving the Metasul LDH™ total hip system. To prevent intra-observer variation the metal ion concentrations was analysed by an approved Central Laboratory. The Central Laboratory provided specimen collection kits for the transfer of blood specimens to the Laboratory for analysis. The Laboratory provided the results to the Investigators. The cobalt and chromium was measured by induced coupled plasma mass spectrometry (ICP-MS). BUN, creatinine and GFR will be determined locally.

SUMMARY:
The Zimmer Hip Resurfacing System Post-Market Clinical Follow-up study will examine the safety and efficacy of this device in the young and/or active patient with advanced hip disease.

DETAILED DESCRIPTION:
This is a multi-center, prospective, non-controlled post market surveillance study. The objective of this study is to obtain survival and outcome data on the Zimmer Hip Resurfacing System. This will be assessed by analysis of standard scoring systems, radiographs and adverse event records. Data will be used to monitor pain, mobility and survivorship, and to confirm the safety and efficacy of the Zimmer Hip Resurfacing System. Serum metal ion levels (cobalt and chromium) will also be collected pre-operatively and again at 6 months, 1 year, 2 years and 5 years. This procedure will offer an option to these patients who would otherwise require and likely outlive a conventional total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Patient selection without bias to race or gender.
2. Patient is ≥ 18 and ≤ 65 years of age.
3. Female patients only, if

   1. Actively practicing a contraceptive method, or
   2. Surgically sterilized, or
   3. Post-menopausal
4. Pre-operative Harris Hip Score ≤ 70.
5. Primary surgical hip candidate, suffering from hip pain and/or disability due to degenerative joint disease (inflammatory or non-inflammatory), based on physical examination and history, which may include the following diagnosis:

   1. Non-inflammatory degenerative joint disease (NIDJD), e.g. avascular necrosis or osteoarthritis
   2. Inflammatory joint disease (IJD), e.g., rheumatoid arthritis
6. Patient is willing and able to cooperate in prescribed post-operative therapy.
7. Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.
8. Patient has participated in the Informed Consent process and has signed an Ethics Committee approved Informed Consent.

Exclusion Criteria:

1. Patient has an acute, chronic, local or systemic infection.
2. Patient is skeletally immature.
3. Patient is known to be pregnant.
4. Patient has a severe muscular, neural or vascular disease that endangers the involved extremity.
5. Patient has an insufficient acetabular or femoral bone stock in which good anchorage of the implants are unlikely or impossible, including, but not limited to:

   1. patient with severe osteopenia,
   2. patients with a family history of severe osteoporosis or osteopenia,
   3. patients with osteonecrosis or avascular necrosis (AVN) with >50% involvement of the femoral head (regardless of FICAT grade), or
   4. patients with local bone tumors and/or cysts of the femoral head > 1 cm
6. Patient has a total or partial absence of the muscular or ligamentous apparatus.
7. Patient has known moderate to severe renal insufficiency.
8. Patient has a known clinical condition which may interfere with the patient's outcome, including but not limited to:

   1. immunocompromised conditions (AIDS),
   2. organ transplant,
   3. high doses of corticosteroids etc
9. Patient is severely overweight (BMI > 40)
10. Patient is scheduled for simultaneous bilateral total hip replacement.
11. OPERATIVE (IPSILATERAL) HIP: Patient has a total prosthetic hip replacement device, surface arthroplasty, endoprosthesis or femoral and/or acetabular osteosynthesis.
12. CONTRALATERAL HIP: Patient has had a hip replacement, surface arthroplasty or endoprosthesis, within the past 12 months, unless previously enrolled in this clinical study.
13. Patient is:

    1. a prisoner,
    2. mentally incompetent,
    3. a known alcohol or drug abuser,
    4. anticipated to be non-compliant
14. Patient has participated in a study of any other investigational device (drug, device or biologic) within the past 12 months. Exception: previous enrollment in the Zimmer Hip Resurfacing clinical study.
15. Patient has a known allergy to one of the constituents of the implant, e.g. cobalt, chromium, nickel, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-08-01 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (1):
- Medizinische Fakultàt Carl Gustav Carus der Technischen Universität Dresden, Dresden, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Who Received Metasul Monoblock in Hip Resurfacing: Patients who received the Zimmer Hip Resurfacing System utilising the Metasul Monoblock Component™ Cup in a Hip Resurfacing Application with the Durom® Hip Resurfacing Femoral Component and whose Serum metal ion levels is being measured.
  Serum Metal ion levels determined to monitor changes in chromium and cobalt levels: Analyses will be performed pre-operatively, 6 months, 1 year, 2 years and 5 years postoperatively for all study subjects enrolled in this study, as well as, all revision study subjects receiving the Metasul® LDH™ total hip system. To prevent intra-observer variation the metal ion concentrations will be analysed by an approved Central Laboratory. The Central Laboratory will provide specimen collection kits for the transfer of blood specimens to the Laboratory for analysis. The Laboratory will provide the results to the Investigators. The cobalt and chromium will be measured by induced coupled plasma mass spectrometry (ICP-MS). BUN, creatinine and GFR will be determined locally.
Period: Overall Study
Arm/Group | Patients Who Received Metasul Monoblock in Hip Resurfacing
Started | 45
Completed | 36
Not Completed | 9
Not completed — Death | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- Patients Who Received the Zimmer Hip Resurfacing System: The Zimmer Hip Resurfacing System is designed for the treatment of degenerative diseases or trauma of the hip. The system is intended to reduce pain and increase hip mobility.
  The Zimmer Hip Resurfacing System may be used for the following indications:
  * Non inflammatory degenerative joint disease (NIDJD), e.g. avascular necrosis, primary osteoarthritis and post traumatic arthritis
  * Inflammatory joint disease (IJD), e.g. rheumatoid arthritis.
Arm/Group | Patients Who Received the Zimmer Hip Resurfacing System
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 50.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 45
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (3.9)
Weight [Mean (Standard Deviation); unit: Kg] | 90.7 (13.0)
Height [Mean (Standard Deviation); unit: Cm] | 178.2 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Implant Survival
Description: The primary endpoint for this study is implant survival at 10 years which is assessed by revision of the Metasul Monoblock Component Cup calculated using the Kaplan-Meier Survival Estimation. The survivorship with Kaplan-Meier (K-M) was calculated at 10 year for endpoint revision of any component.
Time Frame: 10 years post-surgery
Population: All study patients involved in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Patients Who Received Metasul Monoblock in Hip Resurfacing: Patients who received the Zimmer Hip Resurfacing System utilising the Metasul Monoblock Component Cup in a Hip Resurfacing Application with the Durom Hip Resurfacing Femoral Component and whose Serum metal ion levels is being measured.
  Serum Metal ion levels determined to monitor changes in chromium and cobalt levels: Analyses will be performed pre-operatively, 6 months, 1 year, 2 years and 5 years postoperatively for all study subjects enrolled in this study, as well as, all revision study subjects receiving the Metasul LDH™ total hip system. To prevent intra-observer variation the metal ion concentrations will be analysed by an approved Central Laboratory. The Central Laboratory will provide specimen collection kits for the transfer of blood specimens to the Laboratory for analysis. The Laboratory will provide the results to the Investigators. The cobalt and chromium will be measured by induced coupled plasma mass spectrometry (ICP-MS). BUN, creatinine and GFR will be determined locally.
Arm/Group | Patients Who Received Metasul Monoblock in Hip Resurfacing
Number analyzed (Participants) | 45
percentage of participants | 95.39 [82.79 to 98.83]

2. Secondary Outcome: Harris Hip Score
Description: The Harris Hip Score (HHS) is an outcome measure that includes a series of questions answered by the patient and physical examinations recorded by a qualified health care professional. The HHS covers four domains: pain, function and functional activities, absence of deformity and range of motion. The total score vary from a range of 0 - 100. The outcome score can be categorized as Excellent: 90-100; Good: 80-90; Fair: 70-80; Poor: < 70.
Time Frame: Preop, 6 months, 1 year, 2 year, 3 year, 5 year, 7 year and 10 years post-surgery
Population: The mean Harris Hip Score and standard deviation for all study patients is presented in the results section below for all follow up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received Metasul Monoblock in Hip Resurfacing
Number analyzed (Participants) | 45
score on a scale
  Preop: number analyzed (Participants) | 42
  Preop | 55.1 (8.2)
  6 Months: number analyzed (Participants) | 42
  6 Months | 93.9 (7.4)
  1 Year: number analyzed (Participants) | 39
  1 Year | 95.3 (7.3)
  2 Year: number analyzed (Participants) | 35
  2 Year | 97.3 (5.3)
  3 Year: number analyzed (Participants) | 28
  3 Year | 96.6 (10.5)
  5 Year: number analyzed (Participants) | 40
  5 Year | 98.6 (3.2)
  7 Year: number analyzed (Participants) | 40
  7 Year | 98.1 (4.1)
  10 Year: number analyzed (Participants) | 33
  10 Year | 97.2 (5.2)

3. Secondary Outcome: Subject Quality-of-life Determined by the SF-12 Questionnaire (Mental Health and Physical Health)
Description: The SF-12 is a multi-purpose short-form (SF) generic measure of health status. It consists of twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). Mental health-related scales include Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH). Scores ranges from 0 to 100, with higher scores indicating better physical and mental health functioning.
Time Frame: Preop, 6 months, 1 year, 2 year, 3 year, 5 year, 7 year and 10 years post-surgery
Population: The mean and standard deviation for SF-12 physical and mental is presented in the results section below for all follow up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received Metasul Monoblock in Hip Resurfacing
Number analyzed (Participants) | 45
score on a scale
  Preop Mental Health SF12 Score: number analyzed (Participants) | 41
  Preop Mental Health SF12 Score | 49.7 (10.7)
  6 Months Mental Health SF12 Score: number analyzed (Participants) | 42
  6 Months Mental Health SF12 Score | 54.3 (8.9)
  1 Year Mental Health SF12 Score: number analyzed (Participants) | 40
  1 Year Mental Health SF12 Score | 55.1 (6.1)
  2 Year Mental Health SF12 Score: number analyzed (Participants) | 35
  2 Year Mental Health SF12 Score | 55.1 (6.8)
  3 Year Mental Health SF12 Score: number analyzed (Participants) | 34
  3 Year Mental Health SF12 Score | 53.9 (7.8)
  5 Year Mental Health SF12 Score: number analyzed (Participants) | 40
  5 Year Mental Health SF12 Score | 56.1 (5.5)
  7 Year Mental Health SF12 Score: number analyzed (Participants) | 39
  7 Year Mental Health SF12 Score | 55.5 (5.6)
  10 Year Mental Health SF12 Score SF12 Score: number analyzed (Participants) | 36
  10 Year Mental Health SF12 Score SF12 Score | 54.6 (7.7)
  Preop Physical Health SF12 Score SF12 Score: number analyzed (Participants) | 44
  Preop Physical Health SF12 Score SF12 Score | 30.5 (8.8)
  6 Month Physical Health SF12 Score: number analyzed (Participants) | 44
  6 Month Physical Health SF12 Score | 47.8 (7.7)
  1 Year Physical Health SF12 Score: number analyzed (Participants) | 40
  1 Year Physical Health SF12 Score | 49.1 (9.7)
  2 Year Physical Health SF12 Score: number analyzed (Participants) | 39
  2 Year Physical Health SF12 Score | 50.2 (9.2)
  3 Year Physical Health SF12 Score: number analyzed (Participants) | 39
  3 Year Physical Health SF12 Score | 49.2 (10.0)
  5 Year Physical Health SF12 Score: number analyzed (Participants) | 40
  5 Year Physical Health SF12 Score | 50.6 (7.7)
  7 Year Physical Health SF12 Score: number analyzed (Participants) | 38
  7 Year Physical Health SF12 Score | 50.8 (6.8)
  10 Year Physical Health SF12 Score: number analyzed (Participants) | 35
  10 Year Physical Health SF12 Score | 48.7 (9.0)

4. Secondary Outcome: Patient's Activity Level Determined by UCLA Score
Description: The UCLA score was a part of the Patient Activity Questionnaire which ascertains the patient's activity level from 1 (low) to 10 (high) in patients undergoing total hip arthroplasty.
Time Frame: Preop, 6 months, 1 year, 2 year, 3 year, 5 year, 7 year and 10 years post-surgery
Population: The mean and standard deviation for UCLA activity score is presented in the results section below for all follow up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received Metasul Monoblock in Hip Resurfacing
Number analyzed (Participants) | 45
score on a scale
  Preop | 4.9 (2.1)
  6 Month: number analyzed (Participants) | 44
  6 Month | 6.5 (1.7)
  1 Year: number analyzed (Participants) | 42
  1 Year | 6.4 (1.9)
  2 Year: number analyzed (Participants) | 41
  2 Year | 6.8 (1.9)
  3 Year: number analyzed (Participants) | 40
  3 Year | 6.9 (2.1)
  5 Year: number analyzed (Participants) | 40
  5 Year | 7.0 (1.7)
  7 Year: number analyzed (Participants) | 39
  7 Year | 6.7 (2.0)
  10 Year: number analyzed (Participants) | 36
  10 Year | 6.6 (1.9)

5. Secondary Outcome: Radiographic Evaluation
Description: Radiographic parameters evaluated were radiolucencies, osteolysis, hypertrophy, subsidence, cup migration, change in cup angle and change in femoral shaft angle. The radiographs related to any significant radiographic findings reported by an Investigator were also be assessed by an Independent Radiographic Reviewer. The data presented in the outcome measure data table represent the Number of Participants with Abnormal or Significant Findings during the course of the study.
Time Frame: Pre-op, 6 weeks, 1,2,3,5,7 and 10 years post operatively 2, 3, 5, 7 and 10 years post-operatively. 2, 3, 5, 7 and 10 years post-operatively.
Population: The significant radiographic findings reported for all patients during the course of the study is presented in the results section below for all follow up time points of occurrence.
Measure: Number; unit: participants
Arm/Group | Patients Who Received Metasul Monoblock in Hip Resurfacing
Number analyzed (Participants) | 45
participants
  6 Month Stem Radiolucency | 1
  7 Years Osteolysis | 1

6. Secondary Outcome: EuroQol 5 Dimension (EQ-5D)
Description: The EuroQol 5 Dimension (EQ-5D) is a standardized Instrument widely used to measure health status. It is a self reported assessment about the patient's quality of life composed of two parts: a questionnaire and a visual analogue scale (VAS). The questionnaire includes 5 questions referring to mobility, selfcare, daily activities, pain/discomfort, and anxiety/depression. Each question can be answered in five ways, indicating no, slight, moderate, severe problems or inability to complete the task. The EQ-5D-5L score ranges from -0.59 to 1, where 1 is the best possible health state. The Visual Analogue Scale (VAS) is a vertical scale ranges from 100 ('The best health you can imagine') to 0 ('The worst health you can imagine') where the patient reports his/her self-rated health. For this study, the VAS score was not calculated.
Time Frame: Preop, 6 months, 1 year, 2 year, 3 year, 5 year, 7 year and 10 years post-surgery
Population: The mean and standard deviation for EQ-5D is presented in the results section below for all follow up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received Metasul Monoblock in Hip Resurfacing
Number analyzed (Participants) | 45
score on a scale
  PreOp | 0.5 (0.2)
  6 Month: number analyzed (Participants) | 42
  6 Month | 0.8 (0.2)
  1 Year: number analyzed (Participants) | 40
  1 Year | 0.9 (0.1)
  2 Year: number analyzed (Participants) | 40
  2 Year | 0.9 (0.2)
  3 Year: number analyzed (Participants) | 40
  3 Year | 0.9 (0.2)
  5 Year: number analyzed (Participants) | 40
  5 Year | 0.9 (0.1)
  7 Year: number analyzed (Participants) | 40
  7 Year | 0.9 (0.2)
  10 Year: number analyzed (Participants) | 36
  10 Year | 0.8 (0.3)

7. Secondary Outcome: Oxford Hip Score
Description: The Oxford Hip Score (OHS) is a patient-reported outcome measure that was developed to specifically assess the patient's perspective of outcome following THA. The OHS consists of twelve questions covering function and pain associated with the hip. To calculate the total score, each response is scored from 0 (worst outcome) to 4 (best outcome) and the sum of all 12 items is reported with a maximum of 48, representing the best score possible. Scores ranges from 0 to 100 and the outcome score can be categorized as Excellent: > 41; Good: 34 - 41; Fair: 27 - 33; Poor: < 27.
Time Frame: Preop, 6 months, 1 year, 2 year, 3 year, 5 year, 7 year and 10 years post-surgery
Population: The mean and standard deviation for Oxford Hip Score is presented in the results section below for all follow up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received Metasul Monoblock in Hip Resurfacing
Number analyzed (Participants) | 45
score on a scale
  Preop | 21.7 (6.8)
  6 Month: number analyzed (Participants) | 44
  6 Month | 35.3 (12.3)
  1 Year: number analyzed (Participants) | 42
  1 Year | 39.1 (11.8)
  2 Year: number analyzed (Participants) | 41
  2 Year | 44.0 (7.2)
  3 Year: number analyzed (Participants) | 40
  3 Year | 44.6 (6.5)
  5 Year: number analyzed (Participants) | 40
  5 Year | 44.7 (5.6)
  7 Year: number analyzed (Participants) | 40
  7 Year | 45.8 (3.6)
  10 Year: number analyzed (Participants) | 36
  10 Year | 44.9 (4.8)

8. Secondary Outcome: Pain and Functional Performance Based on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: The WOMAC Score is a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip. These set of standardized questions are used by doctors to evaluate the condition of osteoarthritis patients. The WOMAC score was an optional form reported for pain and physical function. The test questions are scored on a scale of 0-4, which correspond to: No pain (0), Mild pain (1), Moderate pain (2), Severe pain (3), and Extreme pain (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain (with higher values representing worse outcomes and lower values representing better outcomes) and 0-68 for Physical Function (with higher values representing better outcomes and lower values representing worse outcomes).
Time Frame: Preop, 6 months, 1 year, 2 year, 3 year, 5 year, 7 year and 10 years post-surgery
Population: The mean and standard deviation for the WOMAC pain and physical function score is presented in the results section below for all follow up time points. The number of participants analyzed is not consistent with the numbers in the participant flow module because the numbers reported in the participant flow module represents the number of patients with these form completed at the subsequent follow up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received Metasul Monoblock in Hip Resurfacing
Number analyzed (Participants) | 44
score on a scale
  Preop WOMAC Pain Score | 9.8 (2.8)
  6 Month WOMAC Pain Score | 1.8 (2.8)
  1 Year WOMAC Pain Score: number analyzed (Participants) | 42
  1 Year WOMAC Pain Score | 1.4 (2.5)
  2 Year WOMAC Pain Score: number analyzed (Participants) | 41
  2 Year WOMAC Pain Score | 1.0 (2.1)
  3 Year WOMAC Pain Score: number analyzed (Participants) | 40
  3 Year WOMAC Pain Score | 1.1 (2.2)
  5 Year WOMAC Pain Score: number analyzed (Participants) | 40
  5 Year WOMAC Pain Score | 1.1 (2.3)
  7 Year WOMAC Pain Score: number analyzed (Participants) | 39
  7 Year WOMAC Pain Score | 0.6 (1.1)
  10 Year WOMAC Pain Score: number analyzed (Participants) | 36
  10 Year WOMAC Pain Score | 1.1 (2.1)
  Preop WOMAC Physical Function Score | 33.4 (11.1)
  6 Month WOMAC Physical Function Score | 8.2 (10.7)
  1 Year WOMAC Physical Function Score: number analyzed (Participants) | 42
  1 Year WOMAC Physical Function Score | 5.9 (8.7)
  2 Year WOMAC Physical Function Score: number analyzed (Participants) | 41
  2 Year WOMAC Physical Function Score | 3.8 (7.2)
  3 Year WOMAC Physical Function Score: number analyzed (Participants) | 40
  3 Year WOMAC Physical Function Score | 5.1 (8.3)
  5 Year WOMAC Physical Function Score: number analyzed (Participants) | 40
  5 Year WOMAC Physical Function Score | 4.7 (8.3)
  7 Year WOMAC Physical Function Score: number analyzed (Participants) | 40
  7 Year WOMAC Physical Function Score | 4.1 (7.3)
  10 Year WOMAC Physical Function Score: number analyzed (Participants) | 36
  10 Year WOMAC Physical Function Score | 5.7 (8.1)

ADVERSE EVENTS:
Time Frame: Operative, 6 months, 1 year, 2 year, 3 year, 5 year, 7 year and 10 years post-surgery
Description: Adverse events were grouped into hip related or general adverse events.
Arm/Group | Patients Who Received Metasul Monoblock in Hip Resurfacing
All-Cause Mortality (participants affected / at risk) | 4/45
Serious Adverse Events (participants affected / at risk) | 3/45
Other Adverse Events (participants affected / at risk) | 17/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Who Received Metasul Monoblock in Hip Resurfacing (N=45)
Femoral Neck Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Emergency hospitalization due to a femoral neck fracture
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Pain dragging into the groin with a walking distance of 500m
Translucency (Musculoskeletal and connective tissue disorders) | 1 (1) — Translucency around the left femoral hip stem
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Who Received Metasul Monoblock in Hip Resurfacing (N=45)
Cardiovascular (Cardiac disorders) | 1 (1) — Circulatory Failure
Dermatological (Skin and subcutaneous tissue disorders) | 1 (2) — Erysipelas left tibia and Erysipalas in sore area.
Endocrine (Endocrine disorders) | 1 (1) — Wide knot in thyroid gland
Gastrointestinal (Gastrointestinal disorders) | 1 (1) — Norovirus
Hematological (General disorders) | 1 (1) — Elevated metal ions
Muscoloskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) — Right knee pain
Pulmonary Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Breathlessness
Thigh Groin Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Groin pain
Other General Complications (General disorders) | 1 (1) — Shoulder surgery
Other General Complications (Surgical and medical procedures) | 1 (1) — Bursitis on right elbow
Other General Complications (Gastrointestinal disorders) | 1 (1) — Intestinal inflammation
Other General Complications (Reproductive system and breast disorders) | 1 (1) — Testicular Hydrocele
Other General Complications (Social circumstances) | 1 (1) — Fall from bycicle
Dermatological (Skin and subcutaneous tissue disorders) | 1 (1) — Excema in wound area
Other General Complications (Skin and subcutaneous tissue disorders) | 1 (1) — Exantherm all over body
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Gluteal and femoral pain on knee joint
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Disc hernia

LIMITATIONS AND CAVEATS:
The study devices were taken off the market in 2013.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-02-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT03681639/Prot_SAP_000.pdf